CLINICAL TRIAL: NCT05104671
Title: Thoracic Manipulation Versus Myofascial Release in Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: manar sameh el taher (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, manar sameh el taher, Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shoulder impingement
Record Dates: First submitted 2021-07-18; First posted 2021-11-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Impingement Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scapular stabilization exercises (Active Comparator): Group I (control group) will receive scapular stabilization exercises.
  Interventions: Other: scapular stabilization exercises.
- Thoracic manipulation. (Experimental): Group II will receive scapular stabilization exercises and thoracic manipulation.
  Interventions: Other: scapular stabilization exercises.; Other: Thoracic manipulation.
- Myofascial release (Experimental): Group III will receive scapular stabilization exercises and myofascial release by instrument assisted soft tissue mobilization techniques.
  Interventions: Other: scapular stabilization exercises.; Other: Myofascial release.

INTERVENTIONS:
Other: scapular stabilization exercises. — General Instructions: For all exercises, perform the retraction of the scapula, without performing the elevation of the shoulders, taking the lower angle of the scapula "back and down".
  The exercise intensity was described as repetitions, sets, and holding time. Commonly, 10-20 repetitions and three to five sets held for 3-10 seconds were performed.and the exercises will be:
  1. towel slide
  2. Scapular Clock:
  3. Scapular Proprioceptive Neuromuscular facilitation:
  4. Inferior Glide.
  5. Scapular Orientation Exercise (SOE):
  6. Protraction and retraction in front of a mirror:
Other: Thoracic manipulation. — • Thoracic Thrust Manipulation: The participants were in high sitting and in prone lying position. The therapist was standing next to the patient in a diagonal stance and also behind the patient during high sitting. Thoracic thrust manipulation demonstrated to manipulate specific thoracic segment mainly mid thoracic.
  Other Names: scapular stabilization exercises
  Arms: Thoracic manipulation.
Other: Myofascial release. — The subject will be treated with IASTM.applied to the pectoral muscles and medial brachium with the subject in supine and the glenohumeral joint(GH). placed in 120 º abduction to place adequate tension on the selected tissues in the style of pectoral tightness test .The IASTM technique was performed for 20 seconds parallel to the muscle fibers followed by 20 seconds perpendicular to the muscle fibers with the instrument held at a 45 º angle to the skin.The same IASTM protocol of 20 seconds parallel to the muscle fibers and 20 seconds perpendicular to the muscle fibers was applied to the posterior cuff musculature of the GH joint with the subject in prone and arms in 90 º abduction and internal rotation draped over the side of the plinth . While in the same position, the technique was applied to the periscapular musculature including the, trapezoids, rhomboids, teres minor, teres major, and latissimus dorsi.
  Other Names: scapular stabilization exercises
  Arms: Myofascial release

SUMMARY:
aims: • To investigate the effect of adding thoracic manipulation vs myofascial release to scapular stabilization exercise on pain intensity.

* To investigate the effect of adding thoracic manipulation vs myofascial release to scapular stabilization exercise on pain pressure threshold.
* To investigate the effect of adding thoracic manipulation vs myofascial release to scapular stabilization exercise on shoulder proprioception.
* To investigate the effect of adding thoracic manipulation vs myofascial release to scapular stabilization exercise on shoulder range of motion(ROM).
* To investigate the effect of adding thoracic manipulation vs myofascial release to scapular stabilization exercise on disability of shoulder and hand questionnaire(DASH).

DETAILED DESCRIPTION:
Various researches have been done on rehabilitation of shoulder impingement by addressing either osseous structure or myofascial structure and found to be effective. But no studies could retrieve to compare these two: myofascial release and thoracic manipulation. (Dash & Deepak, 2020). so in this study we will investigate the effect of adding thoracic manipulation versus myofascial release in patients with shoulder impingement syndrome. we will investigate the effect on each of the following: pain intensity will measure by visual analogue scale.(VAS).

proprioception of the shoulder by isokinetic dynamometer. pain pressure threshold by algometer. function by DASH questionnaire and finally ROM by kinovea software.

The subjects will be arranged into three groups: Group I (control group) will receive scapular stabilization exercises.

* Group II will receive scapular stabilization exercises and thoracic manipulation combined with shoulder mobilization.
* Group III will receive scapular stabilization exercises and myofascial release by instrument assisted soft tissue mobilization techniques(IASTM).

the measurements will take before and after treatment programs and after one month of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty patients with shoulder impingement syndrome from both genders their age will be ranged and divided into three groups from 25-40 years.
2. History of shoulder pain for at least one month.
3. Positive Neer's impingement test and Hawkins's kiennedy test.
4. Presence of thoracic hypomobility from clinical evaluation.
5. Provocation of pain above 60 degrees of flexion and abduction.
6. Palpable trigger points on shoulder muscles.

Exclusion Criteria:

1. History of Shoulder girdle fracture, dislocation and surgery
2. Diagnosed with frozen shoulder or rotator cuff tear
3. History of cervicobrachial pain
4. Any neuromuscular pain in upper limb and use of corticosteroids or pain subsiding medication

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Pain in shoulder movement | change from max pain point at 2 months
  will be measured by Visual analog scale(VAS). It consists of a line, often 10 cm long(100mm); its ends are generally labelled with verbal pain anchors (e.g., "no pain" and "pain as bad as it could be"). Patients are asked to indicate the point along the line that best reflects their pain intensity. The majority of the studies showed that visual analogue scale is a valid and reliable scale. Also, it is an interval scale. So, in clinical practice we can use this scale in case of pain measurement as an outcome measure tool.
shoulder function | change from limitation of function at 2 months
  by DASH is a reliable and valid tool for the assessment of shoulder pain and disability in both clinical practice and research.
Shoulder Proprioception (joint of position error) | change from poor proprioception at 2 months
  will be measured by isokinetic dynamometer. Isokinetic dynamometry is considered a valid instrument for assessing muscle strength, and it is often used as a reference standard for other strength assessments.

SECONDARY OUTCOMES:
Shoulder ROM | change from limitation in shoulder ROM at 2 months
  will be measured by Kinovea. Kinovea is a free software used for the analysis, comparison, and evaluation of sports and training. it is a reliable tool for measuring shoulder flexion, abduction, and Internal rotation&external rotation in healthy individuals. Thus, it could be used as a simple alternative to universal goniometry.
Pain pressure threshold in shoulder muscles | change from baseline pain pressure threshold at 2 months
  that Pressure algometer is a worthwhile tool in the diagnosis and treatment evaluation of different orthopedic disorders. . Three consecutive Pressure pain threshold measurements were taken at each point with 20 s rest between measurements, and the mean of the three trials will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Undecided